CLINICAL TRIAL: NCT02435368
Title: The Mechanisms and Significances of Synergistic Effects of Mycophenolic Acid and Lipopolysaccharide on Interleukin-1β Secretion by Mononuclear
Brief Title: The Mechanisms and Significances of Synergistic Effects of Mycophenolic Acid and LPS on IL-1β Secretion by Mononuclear
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The Third Affiliated Hospital of Southern Medical University (Other Government)
Responsible Party: Principal Investigator, Xuechan Huang, Dr.Xuechan Huang, The Third Affiliated Hospital of Southern Medical University
Other Study IDs: 201501001
Record Dates: First submitted 2015-04-25; First posted 2015-05-06 (Estimated); Last update posted 2015-05-06 (Estimated); Status verified 2015-04

CONDITIONS: Lupus Nephritis
MeSH Terms: conditions — Lupus Nephritis | interventions — Mycophenolic Acid

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Peripheral blood was obtained from healthy donors,mononuclear cells (PBMCs) were isolated using Ficoll density gradient centrifugation, and LPS (1 μg/ml) and/or MPA were added. After 12 hours, the supernatants were harvested and stored at -80°C for ELISA.
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: mycophenolic acid — Monocytes were co-cultured with LPS and/or MPA.After 12 hours, the supernatants were harvested and stored at -80°C for ELISA.
  Other Names: mycophenolate mofetil

SUMMARY:
To determine the mechanisms and significances of synergistic effects of mycophenolic acid and LPS on IL-1β secretion by mononuclear

DETAILED DESCRIPTION:
Mycophenolate mofetil (MMF), which inhibits T and B lymphocyte proliferation, is widely used to treat a variety of autoimmune diseases, such as systemic lupus erythematosus (SLE) and lupus nephritis (LN). We are the first to show that mycophenolic acid (MPA), the active metabolite of MMF, in association with lipopolysaccharide (LPS), is able to promote the secretion of interleukin (IL)-1β, which contradicts the traditional conception that immunosuppressants inhibit the secretion of inflammatory factors.

In this study, we first determined the effects of MPA in association with LPS on IL-1β production. Then, we explored whether the synergized effect on IL-1β production was mediated through the nuclear factor （NF）-κB pathway that produces more pro-IL-1β, or through the triggering of NLRP3 inflammasome that leads to enhanced activation of caspase-1 and accelerated degradation of pro-IL-1β into mature IL-1β.

This study is not only conducive to clarify the mechanisms, signal transduction pathways and potential clinical significances of IL-1β production in LPS and MPA combined treatment, but also to provide experimental data as well as theoretical rationales for more effective and more logical immunosuppressive protocols.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Volunteers，age 18-60.

Exclusion Criteria:

* Don't agree with informed consent

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy Volunteers,age 18-60.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2015-04; Primary Completion 2015-11 (Estimated); Study Completion 2016-03 (Estimated)

PRIMARY OUTCOMES:
mean ± SD of percentage of IL-1β production induced by Lipopolysaccharide in associate with MPA in monocytes. | six months

CONTACTS AND LOCATIONS:
Overall Officials: erwei Sun, doctor, Study Director — Third Affiliated Hospital of Southern Medical University
Locations (1):
- Third Affiliated Hospital of Southern Medical University, Guangzhou, Guangdong, China